## STATISTICAL ANALYSIS PLAN

**Study Title:** Efficacy, Safety, and Tolerability of GLS-1200 Topical

Nasal Spray in the Prevention of Incident Confirmed SARS-

CoV-2 Infection

Name of Test Drug: GLS-1200

**Study Number:** T2R-002

**Protocol Version:** 7.0

**Protocol Date:** 26 February 2021

**Analysis Plan Version:** 2.0

**Analysis Plan Date:** 21 January 2022

Analysis Plan Author: Catalyst Clinical Research, LLC

## CONFIDENTIAL AND PROPRIETARY INFORMATION

### SIGNATURE PAGE



21-Jan-2022

Date

GeneOne Life Science Inc.

DocuSigned by:

Susan E. Spruill

Signer Name: Susan E. Spruill

Signing Reason: I approve this document Signing Time: 21-Jan-2022 | 4:07:34 PM CST 6B44CB45B7954FD5B700ED25E98AB084

21-Jan-2022

Signature Date

Susan E. Spruill, MS, PStat®

Statisticial Consultant

**Applied Statistics and Consulting** 

DocuSigned by:

Ahmed Tarig

Signer Name: Ahmed Tariq

Signing Reason: I approve this document Signing Time: 21-Jan-2022 | 2:48:35 PM EST

8A9AFFC7511B48049134C7E9728C3D84

21-Jan-2022

Signature Date

Ahmed Tariq, MS

Biostatistician

Catalyst Clinical Research, LLC

| LIS | Г ОГ АВ | BBREVIATIONS | 5 |
|---|---|---|---|
| 1. | INTRO | DDUCTION | 6 |
| 2. | STUDY | Y OBJECTIVES | 6 |
| | 2.1.<br>2.2.<br>2.3. | Primary Objectives | 6 |
| 3. | STUDY | Y DESIGN AND PLAN | 6 |
| 4. | DETER | RMINATION OF SAMPLE SIZE | 9 |
| 5. | GENEF | RAL ANALYSIS CONSIDERATIONS | 9 |
| 6. | ANAL' | YSIS POPULATIONS | 9 |
| | 6.1.<br>6.2.<br>6.3. | Intent-to-treat (ITT) Population Safety Population Per-protocol (PP) Population | 9 |
| 7. | | Y POPULATION | |
| 8. | 8.1. | Subject Disposition Protocol Deviations Demographics and Baseline Characteristics Medical History Prior and Concomitant Medications Drug Exposure Treatment Compliance ACY ANALYSES Definition of the Primary Efficacy Endpoint | 91010101011 |
| | 8.2.<br>8.3.<br>8.4.<br>8.5.<br>8.6. | Analysis of the Primary Efficacy Endpoint Definition of the Secondary Efficacy Endpoint Analysis of the Secondary Efficacy Endpoint Definition of the Exploratory Efficacy Endpoint Analysis of the Exploratory Efficacy Endpoint | 11<br>11<br>12 |
| 9. | SAFET | ΓΥ ANALYSES | 12 |
| | 9.1. | Adverse Events 9.1.1. Severity 9.1.2. Relationship 9.1.3. Serious Adverse Events 9.1.4. Treatment-Emergent Adverse Events (TEAEs) 9.1.4.1. Definition of Treatment-Emergent 9.1.4.2. Incomplete Dates | |
| | 9.2.<br>9.3.<br>9.4. | 9.1.5. Summaries of Adverse Events. Clinical Laboratory Evaluations. Vital Signs. ECG Results. Physical Evam | 14<br>14<br>14 |

| APPENDIX A: PRESENTATION OF DATA AND PROGRAMMING SPECIFICATIONS | 16 |
|-------------------------------------------------------------------|----|
| APPENDIX B: TABLE OF CONTENTS FOR STATISTICAL TABLES AND LISTINGS | 19 |
| APPENDIX C: TABLE LAYOUTS | 23 |
| APPENDIX D: FIGURE LAYOUTS | 47 |
| APPENDIX E: LISTING LAYOUTS | 50 |

### LIST OF ABBREVIATIONS

AΕ adverse event

ATC **Anatomical Therapeutic Chemical** 

BMI body mass index beats per minute bpm case report form **CRF** Clinical Study Report **CSR DBP** diastolic blood pressure electrocardiogram **ECG** 

early termination Food and Drug Administration FDA

GI gastrointestinal

EΤ

hepatitis B surface antigen HBsAg

hepatitis C virus **HCV** 

International Conference on Harmonisation ICH

ΙP **Investigational Product** 

ITT Intent-to-Treat

MedDRA Medical Dictionary for Regulatory Activities

OTC over-the-counter PT preferred term SAE serious adverse event SBP systolic blood pressure

standard deviation SD SOC system organ class

tables, figures, and listings **TFLs** ULN upper limit of normal World Health Organization WHO

#### 1. INTRODUCTION

This document outlines the statistical methods to be implemented during the analyses of data collected within the scope of GeneOne Life Science Inc.'s Protocol T2R-002 [Efficacy, Safety, and Tolerability of GLS-1200 Topical Nasal Spray in the Prevention of Incident Confirmed SARS-CoV-2 Infection]. The purpose of this plan is to provide specific guidelines from which the statistical analyses will proceed. Any deviations from this plan will be documented in the clinical study report (CSR).

The reader is referred to the following complementary documents:

- Protocol T2R-002, version 7.0, dated 26Feb2021
- Case Report Form (CRF), version 1.017, dated 04Jun2020
- Symptom Diary, version 2, dated 16Apr2020
- Treatment Diary, version 1, dated 28 Mar2020
- DMP, version 1.0, dated 19Jun2020

#### 2. STUDY OBJECTIVES

# 2.1. Primary Objectives

The primary objectives of the study are to evaluate the safety and tolerability of GLS-1200 topical nasal spray as well as the incidence in the diagnosis of PCR-confirmed SARS-CoV-2 infection by treatment group.

# 2.2. Secondary Objective

The secondary objective is to assess the documentation of symptoms consistent with SARS-CoV-2 infections relative to treatment group.

# 2.3. Exploratory Objective

The exploratory objective of the study is to assess the incidence of seroconversion in serum and the relationship of taste receptor genetics to incidence of SARS-CoV-2 infection relative to treatment group.

#### 3. STUDY DESIGN AND PLAN

This is a Phase II, placebo-controlled, double-blind study of GLS-1200 topical nasal spray to assess the safety, tolerability, and ability to reduce the incidence of confirmed SARS-CoV-2 infection. Following recruitment and informed consent, those meeting enrollment criteria will be randomized 2:1 (GLS-1200:Placebo). Participants will initiate topical nasal spray applications immediately after randomization and will continue for 4 weeks. Participants will self-administer drug three times daily. Follow-up will continue through 6 weeks since some cases of SARS-CoV-2 infection may not be apparent until after the primary treatment period has concluded. The primary outcome measurements are safety, tolerability, and reduction in the diagnosis of PCR-confirmed SARS-CoV-2 infection. Secondary measures will assess the incidence of symptoms

between each visit, by treatment group. In addition the average number of days subjects experience each symptom will be summarized by treatment group. Exploratory measures will assess the incidence of seroconversion in serum and the relationship of taste receptor genetics to incidence of SARS-CoV-2 infection both relative to treatment group.

**Table 1: Schedule of Assessments** 

| Tests and Observations | Day 0 | Week 2 | Week 4 | Week 6 | Unscheduled |
|---|---|---|---|---|---|
| Permitted window (days) | | ±3d | ±3d | ±3d | N/A |
| Clinical Evaluations | | | | | |
| Obtain Written Informed Consent | X | | | | |
| Confirm Eligibility Criteria | X | | | | |
| Demographics | X | | | | |
| Medical History and Concomitant Medications | X | X | X | X | |
| Physical Exam, height, weight, and Vital Signs <sup>1</sup> | X | X | X | X | X |
| Safety Evaluations | | | | | |
| Record Adverse Events | | X | X | X | X |
| Provide participant diary | X | | | | |
| Collect and review participant diary | | $X^2$ | X | X | |
| Perform 12-lead ECG | X | | X | | |
| Pregnancy test <sup>3</sup> | X | X | X | | |
| Blood for Hematology: CBC with differential | X | | X | | |
| Blood for Chemistry: Sodium, potassium, bicarbonate, glucose, BUN, Cr | X | | X | | |
| Study Related Procedures | | | • | | |
| Dispense study drug & device, provide training | X | | | | |
| Collect nasopharyngeal swabs for viral PCR | X | X | X | X | X |
| Collect serum for viral antibodies | X | X | X | X | |
| Collect plasma for measurement of quinine | | X | | | |
| Collect saliva for TAS2R genotyping | X | | | | |
| Estimated Blood Volume per Visit (mL) | 40 | 25 | 40 | 20 | |

<sup>&</sup>lt;sup>1</sup> A targeted physical exam will be performed at Weeks 2, 4 and 6 and at unscheduled visits.

<sup>2</sup> The participant diary will only be reviewed at Weeks 2 and 4; it will be reviewed and collected at Week 6.

<sup>3</sup> A urine pregnancy test will be administered.

#### 4. DETERMINATION OF SAMPLE SIZE

The sample size for this study assumes an infection rate in the placebo group of 10%. A 2:1 randomization of 225 subjects would have a power of 80.8% to detect a difference of 9% between groups at alpha = 0.05 assuming 1% of individuals in the treatment group are confirmed to be infected with SARS-CoV-2.

#### 5. GENERAL ANALYSIS CONSIDERATIONS

The statistical analysis results will be reported using tables, listings, and figures (TLFs). Summaries of continuous variables will display means, standard deviations (SDs), medians, minimums, maximums and the number of observations. Summaries of categorical variables will display frequency counts and percentages.

All analyses will be performed using SAS® Version 9.4 or higher.

#### 6. ANALYSIS POPULATIONS

## 6.1. Intent-to-treat (ITT) Population

The ITT Population will include all randomized to treatment allocation.

# 6.2. Safety Population

The Safety Population will include all subjects who received at least one dose of study treatment.

# 6.3. Per-protocol (PP) Population

The PP Population will include all subjects who complete the trial and who receive  $\geq$  90% of the study treatments through to either diagnosis of SARS-CoV-2 infection (study end point) or to end of study (4 weeks), based on subject's completed doses on the treatment diary form, and who have no significant protocol deviations.

#### 7. STUDY POPULATION

#### 7.1. Subject Disposition

The number and percentage of subjects in each analysis population, who completed the study and who discontinued prior to study completion will be presented by treatment (GLS-1200 and placebo) and overall. Disposition will also by summarized by site. Subjects who discontinued prior to completing the study will also be summarized by reason for discontinuation.

Subject disposition will also be listed.

#### 7.2. Protocol Deviations

Protocol deviations with significance will be listed.

# 7.3. Demographics and Baseline Characteristics

Demographics, baseline data, vital signs, medical history, prior and concomitant medications and treatments will be summarized by means of descriptive statistics: continuous variables as mean, median, SD, minimum/maximum ranges and categorical variables as frequencies and percentages, stratified by treatment arms and overall, based on the ITT population. These summaries will also by provided by site. Demographic and baseline characteristics will be listed.

# 7.4. Medical History

Medical history verbatim terms collected from the CRF will be mapped to system organ classes (SOCs) and preferred terms (PTs) using the Medical Dictionary for Regulatory Activities (MedDRA) (version 23.0).

Summaries (number and percentage of subjects) of medical history by SOC and PT will be provided by treatment and overall.

A listing of medical history will be provided.

#### 7.5. Prior and Concomitant Medications

Medication verbatim names collected from the CRF will be mapped to Anatomical Therapeutic Chemical (ATC) Classes and Preferred Names using the World Health Organization's WHODrug Global March 2020 version. Preferred Names will consist of only the base compounds and not the salts (e.g., Naproxen Sodium will be listed only as Naproxen). Concomitant medications will be summarized for each treatment by ATC class and preferred name. Prior and concomitant medications will be listed.

A prior medication is defined as a medication that was administered up to 8 weeks prior to first dose of study treatment. All other medications will be considered concomitant.

## 7.6. Drug Exposure

Exposure summaries of duration of exposure, total number of doses taken, and total number of doses missed, will be provided by treatment. Duration of exposure is defined as the date of last dose minus the date of first dose, regardless if any doses were missed in between.

Dosing data collected from treatment diaries will be listed along with any treatment side effects or device issues, and the number of known or suspected exposures to SARS-CoV-2.

# 7.7. Treatment Compliance

Treatment compliance is defined as the total number of administered doses, as recorded in the treatment diary, divided by the total number of planned doses. Each recorded dose will be considered to be a complete dose of study drug. Descriptive statistics of treatment compliance as well as the proportion of subjects falling into different treatment compliance categories (<50%, 50%-80%, and >80%) will be summarized by treatment group.

Unless differences are observed between sites in the baseline characteristics and demographics that would confound interpretation of efficacy and safety results, all efficacy and safety will be summarized over both sites. If there are concerns for confounded results due to site differences in demographic or baseline characteristics, then all efficacy and safety results will be subset by sites as well as overall. However, no treatment comparisons within sites will be made since the study is not powered to assess treatment effect within sites.

#### 8. EFFICACY ANALYSES

# 8.1. Definition of the Primary Efficacy Endpoint

The primary efficacy endpoint is the incidence of SARS-CoV-2 infection, confirmed by PCR at any time within four weeks of treatment initiation. Participants will be queried as to any new diagnosis of SARS-CoV-2 infection, defined as a positive PCR test for SARS-CoV-2. Subjects who test negative for SARS-CoV-2 infection at Weeks 2 and 4 will be considered treatment successes. Subjects who are lost to follow-up, require rescue therapy, discontinue the study prior to completion of Week 4, or test positive for SARS-CoV-2 infection at at any point within four weeks of treatment initiation will be considered treatment failures. All deaths will be considered as treatment failures.

### 8.2. Analysis of the Primary Efficacy Endpoint

The number and percentage of treatment failures as well as treatment successes will be presented by treatment and compared using Fisher's exact test. Additionally, the number and percentage of subjects who test positive as well as those who test negative for SARS-CoV-2 infection will be provided by treatment at each visit (Weeks 2, 4 and 6). This summary and analysis will be performed for both the ITT and PP populations.

## 8.3. Definition of the Secondary Efficacy Endpoint

The secondary efficacy endpoint is the documentation of symptoms consistent with SARS-CoV-2 infections. Subjects will be instructed to maintain a symptom diary that includes those symptoms considered common for SARS-CoV-2. The diary is inclusive of symptoms identified by the World Health Organization for a diagnosis of SARS-CoV-2 as well as more recently identified symptoms such as conjunctivitis, diarrhea, and loss of taste or smell. Each symptom will be scored as present (score of 1) or absent (score of 0) and will be recorded in the symptom diary on a daily basis.

# 8.4. Analysis of the Secondary Efficacy Endpoint

The incidence of each symptom will be summarized by treatment group for each two week interval. In addition, the average number of days subjects had each symptom throughout the study period (6 weeks) will be summarized by treatment group. Summaries will be presented noncumulatively by visit as well as cumulatively over 4 weeks of treatment. The secondary analysis will be performed for the ITT population.

# 8.5. Definition of the Exploratory Efficacy Endpoint

The exploratory efficacy endpoint is the incidence of SARS-CoV-2 seroconversion.

# 8.6. Analysis of the Exploratory Efficacy Endpoint

The cumulative number and percentage of subjects who seroconvert at each post-baseline visit will be presented by treatment for the ITT population. The relationship of taste receptor genetics to incidence of SARS-CoV-2 infection relative to treatment group will be examined on an adhoc basis and is outside the scope of this document.

#### 9. SAFETY ANALYSES

All safety analyses will be based on the Safety Population.

#### 9.1. Adverse Events

An adverse event (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body, or worsening of a pre-existing condition, temporally associated with the use of a product whether or not considered related to the use of the product. In this study, such changes will be monitored, classified, and summarized, as Clinical or Laboratory AEs. Medical conditions/diseases present before starting the investigational drug will be considered adverse events only if they worsen after starting study treatment. Verbatim terms on CRFs will be mapped to preferred terms (PTs) and system organ classes (SOCs) using the Medical Dictionary for Regulatory Activities (MedDRA) (version 23.0).

# **9.1.1.** Severity

AEs are graded by the investigator as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (potentially life threatening) or Grade 5 (death) according to the NCI Common Terminology Criteria for Adverse Events version 5.0.

## 9.1.2. Relationship

Based on the criteria described below, AEs will be classified according to one of the following categories:

- Related the investigator considers that there is a causal relationship between the event and study drug
- Probably related the investigator considers that there is a probability of a causal relationship of the event to the study drug
- Possibly related the investigator considers that there is a possible causal relationship of the event to the study drug
- Unlikely related the investigator considers that there is an unlikely causal relationship of the event to the study drug
- Not related the investigator considers that the event has no relationship to administration of the study drug

For the purpose of analysis, related AEs are those reported as "Related," "Probably related," "Possibly related" and unrelated AEs are those reported as "Unlikely related" or "Not related." Events for which the investigator did not record relationship will be considered related for analysis. Data listings will show relationship as missing.

#### 9.1.3. Serious Adverse Events

An SAE is any adverse drug experience occurring at any dose that results in any of the following outcomes:

- Death during the period of surveillance defined by the protocol;
- Is immediately life-threatening (e.g., participant was, in the view of the Investigator, at immediate risk of death from the event as it occurred). This does not include an AE that, had it occurred in a more serious form, might have caused death;
- An event requiring inpatient hospitalization or prolongation of existing hospitalization during the period of protocol defined surveillance (including any overnight stay in the hospital, regardless of the length of stay, even if the hospitalization is only a precautionary measure to allow continued observation. However, hospitalization (including hospitalization for an elective procedure) for continued treatment or assessment of a pre-existing condition that has not worsened, does not constitute an SAE. NOTE: Evaluation in a physician's office, or at a hospital or other urgent care setting in an observational, non-admitted status regardless of the time period of observation, does not constitute an SAE;
- Results in congenital anomaly or birth defect;
- Results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions;
- Is an important medical event that may not result in death, be life threatening, or require hospitalization, but based upon appropriate medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed above. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization;
- Is medically significant or requires intervention to prevent one or other of the outcomes listed above.

## 9.1.4. Treatment-Emergent Adverse Events (TEAEs)

#### 9.1.4.1. Definition of Treatment-Emergent

TEAEs are events that either:

a) began on or after the date and time of first dose or

CONFIDENTIAL Page 13 21JAN2022

b) had no recorded start date and the stop date is not before the date and time of first dose.

### 9.1.4.2. Incomplete Dates

If the date of onset is incomplete, then the month and year (or year alone if month is not recorded) of onset determine treatment emergence as follows. The event is treatment emergent if the month and year of onset (or year of onset) of the event is the same as or after the month and year (or year) of date of first dose.

#### 9.1.5. Summaries of Adverse Events

An overall summary of AEs will display, by treatment, the number and percentage (with 95% exact binomial confidence interval) of subjects who had any TEAE, whose strongest TEAE relationship to study drug is related or not related, whose maximum TEAE severity is mild, moderate, or severe, who had any SAE, any Serious TEAE, any TEAE leading to study discontinuation, and any TEAE leading to death.

The following summaries (number and percentage of subjects) of AEs (by SOC and PT) will be provided by treatment:

- All TEAEs
- All TEAEs by strongest relationship
- All TEAEs by maximum severity grade
- All Serious AEs
- All Serious TEAEs
- All TEAEs leading to study discontinuation
- All TEAEs leading to death

These summaries will present the number and percentage of subjects with at least one qualifying AE. Subjects may have more than one AE per SOC and PT. Each summary will be ordered by descending order of incidence of SOC and PT within each SOC.

In addition to the by-treatment summaries, data listings will be provided for the following:

- All AEs (with a flag indicating whether the event is treatment emergent)
- SAEs
- AEs leading to study discontinuation
- Deaths

# 9.2. Clinical Laboratory Evaluations

Shift from baseline in laboratory parameter results (indicated as Low, Normal, or High) will be summarized for each post-baseline visit. Mean (+/- SD) laboratory parameter values will be graphically presented over time by treatment. All laboratory parameters will be listed and include indicators for low/high and clinical significance as determined by the investigator.

# 9.3. Vital Signs

Vital signs (temperature, heart rate, systolic blood pressure (SBP), diastolic blood pressure (DBP)) will be summarized using descriptive statistics (sample size, mean, SD, median, minimum, and maximum) at baseline and at each post-baseline time point by treatment. Change from baseline will also be summarized at each post-baseline time point. Mean (+/- SD) Vital Sign values will be graphically presented over time by treatment. All vital signs results will be listed.

#### 9.4. ECG Results

Shift from baseline in 12-Lead ECG overall interpretion (results are Normal, Abnormal Not Clinically Significant (NCS), or Abnormal Clinically Significant (CS)) will be summarized at each post-baseline visit by treatment. Mean (+/- SD) continuous ECG parameter values will be graphically presented over time by treatment.

Additionally, the number and percentage of subjects will be summarized for the following QTcF Interval result categories at baseline and each post-baseline visit by treatment:

- <=450 msec (males) or <=470 msec (females)
- >450 msec (males) or >470 msec (females)
- Change from baseline <=60 msec (only applies to Week 4)
- Change from baseline >60 msec (only applies to Week 4)

A listing of ECG results will present the interpretations of abnormalities and whether these are considered clinically significant by the investigator.

# 9.5. Physical Exam

Physical exam findings will be listed.

#### APPENDIX A: PRESENTATION OF DATA AND PROGRAMMING SPECIFICATIONS

#### **Tables**

- Formal organization of tabulations may be changed during programming if appropriate, e.g., tables for the different variables may be combined into a single table, or tables with more than one variable may be split into several tables.
- Means, medians, and quartiles will be presented to one more decimal place than the raw data. SDs will be presented to two more decimal places than the raw data. Minimums and maximums will be reported with the same number of decimal places as the raw data.
- Percentages will be presented to the tenths place.
- For frequency counts of categorical variables, categories whose counts are zero will be displayed for the sake of completeness. For example, if none of the subjects discontinue due to "lost to follow-up," this reason will be included in the table with a count of 0. Categories with zero counts will not have zero percentages displayed.
- The last footnote will be "Reference: xxx", where xxx indicates the source listing number(s).

## Listings

- Formal organization of the listing may be changed during programming if appropriate, e.g., additional variables may be included, change in the column order, or the listing may be split into multiple parts due to space constraints, etc.
- If not otherwise specified, all data listings will be sorted by treatment, subject number, visit, and date/time as appropriate.
- All date values will be presented in a ISO 8601 date (e.g., 2001-08-29) format.
- All observed time values will be presented using a 24-hour clock HH:MM:SS format (e.g., 01:35:45 or 11:26). Seconds will only be reported if they were measured as part of the study.

#### Missing or incomplete dates, i.e., AEs and concomitant medications

The most conservative approach will be systematically considered. If the AE onset date is missing or incomplete, it is assumed to have occurred during the study treatment phase (i.e., considered a TEAE) except if the partial onset date or other data such as the stop date, indicates differently. Similarly, a medication with partial start and stop dates could be considered as a concomitant treatment.

The following algorithms will be applied to missing and incomplete start and stop dates:

#### **Start Dates**

- If the day portion of the start date is missing, then the start date will be estimated to be equal to the date of IP administration, provided the start month and year are the same as IP administration and the stop date is either after IP administration or completely missing. Otherwise, the missing day portion will be estimated as '01'.
- If both the day and month portions of the start date are missing, then the start date will be estimated to be equal to the date of IP administration, provided the start year is the same as IP administration and the stop date is either after IP administration or completely

missing. Otherwise, the event will be assumed to start on the first day of the given year, e.g., 2013-??-?? is estimated as 2013-01-01.

- If the start date is completely missing and the stop date is either after IP administration or completely missing, the start date will be estimated to be the day of IP administration. Otherwise, the start date will be estimated to be the first day of the same year as the stop date. All other non-AE and non-concomitant medication day calculations where only partial dates are available will be handled as follows: the first day of the month will be used in the calculations if the day part of a start date is missing while January 1 will be employed if both the month and day parts of a start date are missing.
- For treatment start dates, if patients are randomized and have non-missing visit data for Week 4 as well as non-missing treatment diary data, then start date is set to earliest treatment diary date. If patient's treatment diary data is missing or Week 4 visit is missing, then treatment start date is set to earliest recorded exposure date. Drug dispensation date is used as treatment start date if no other data is available.

# **Stop Dates**

- If only the day of resolution is unknown, the day will be assumed to be the last of the month, e.g., 2013-01-?? will be treated as 2013-01-31.
- If both the day and month of resolution are unknown, the event will be assumed to have ceased on the last day of the year, e.g., 2013-??-?? will be treated as 2013-12-31.
- If the stop date is completely missing or the event is continuing, the event will be assumed to be after IP administration and will be left as missing.
- For treatment stop dates, if patient has non-missing treatment diary data but has data gaps of more than 3 days, then treatment stop date is set to start date + 28 days. If treatment diary data is non-missing and there are no data gaps of 3 days or more then treatment stop date is set to last treatment diary date. If treatment diary data is missing but patient is recorded to have completed study, then treatment stop date is set to start date + 28 days. Finally, if treatment diary data is missing and patient has not completed the study, then treatment stop date is set to study withdrawal date.

#### **Standard Calculations**

Variables requiring calculation will be derived using the following formulas:

- Study Day The day in relation to the first dose date (Day 0), calculated as date first dose date.
- Days A duration expressed in days between two dates (start date and end date) is calculated using the formulas noted below:
- duration in days = end date start date + 1, where end date  $\ge$  start date
- duration in days = end date start date, where end date < start date

- Months A duration expressed in months is calculated as the number days divided by 365.25/12 (~30.4).
- Years A duration expressed in years between one date (date1) and another later date (date2) is calculated using the formula: duration in years =  $\frac{\text{date2-date1+1}}{365.25}$
- Height Height entries made in inches (in) are converted to centimeters (cm) using the following formula: height (cm) = height (in)  $\times$  2.54
- Weight Weight entries made in pounds (lb.) are converted to kilograms (kg) using the following formula: weight (kg) = weight (lb.) / 2.2046
- Temperature Temperature entries in degrees Fahrenheit are converted to degrees centigrade using the following formula: temp (degrees centigrade) = 5/9 × [temp (degrees Fahrenheit) 32]
- Change from baseline Change from baseline will be calculated as: Change = post baseline value baseline value
- Percent change from baseline Change from baseline will be calculated as: percent change from baseline = [(post baseline value baseline value) / baseline value]
   × 100

## APPENDIX B: TABLE OF CONTENTS FOR STATISTICAL TABLES AND LISTINGS

The following TL numbering is completed according to ICH guidelines. The ICH heading number and description are in **bold**. Minor changes from this planned index do not need to be amended in the SAP. Formal organization of tabulations may be changed during programming if appropriate, e.g., tables for the different variables may be combined into a single table, or tables with more than one variable may be split into several tables.

## **List of Tables**

| ICH | Table | |
|---|---|---|
| Heading | Number | Table Description |
| 14.1 | | DEMOGRAPHIC/BASELINE DATA |
| | 14.1.1.1 | Subject Disposition (All Subjects) |
| | 14.1.1.2 | Reason For Screen Failure (All Screen Failure Subjects) |
| | 14.1.2 | Demographic and Baseline Characteristics (Safety Population) |
| | 14.1.3 | Medical History (Safety Population) |
| | 14.1.4 | Concomitant Medications (Safety Population) |
| | 14.1.5 | Exposure and Treatment Compliance (Safety Population) |
| 14.2 | | EFFICACY DATA |
| | 14.2.1.1 | Incidence of SARS-CoV-2 Infection by Visit (ITT Population) |
| | 14.2.1.2 | Incidence of SARS-CoV-2 Infection by Visit (PP Population) |
| | 14.2.2 | Incidence of Individual Symptoms and Average Number of Days |
| | | with Symptoms by Visit Interval (ITT Population) |
| | 14.2.3 | Cumulative Incidence of SARS-CoV-2 Seroconversion by Visit |
| | | (ITT Population) |
| 14.3 | | SAFETY DATA |
| 14.3.1 | | Displays of Adverse Events |
| | 14.3.1.1 | Overall Summary of Adverse Events (Safety Population) |
| | 14.3.1.2 | Treatment-Emergent Adverse Events by System Organ Class and |
| | | Preferred Term (Safety Population) |
| | 14.3.1.3 | Treatment-Emergent Adverse Events by System Organ Class, |
| | | Preferred Term, and Strongest Relationship to Study Drug (Safety |
| | | Population) |
| | 14.3.1.4 | Treatment-Emergent Adverse Events by System Organ Class, |
| | | Preferred Term, and Maximum Severity Grade (Safety Population) |
| | 14.3.1.5 | Related Treatment-Emergent Adverse Events by System Organ |
| | | Class, Preferred Term, and Maximum Severity Grade (Safety |
| | | Population) |
| 14.3.2 | | Serious and Significant Adverse Events |
| | 14.3.2.1 | Serious Adverse Events by System Organ Class and Preferred |
| | | Term (Safety Population) |
| | 14.3.2.2 | Serious Treatment-Emergent Adverse Events by System Organ |
| | | Class and Preferred Term (Safety Population) |

| ICH | Table | |
|---|---|---|
| Heading | Number | Table Description |
| | 14.3.2.3 | Treatment-Emergent Adverse Events Leading to Study |
| | | Discontinuation by System Organ Class and Preferred Term |
| | | (Safety Population) |
| | 14.3.2.4 | Treatment-Emergent Adverse Events Leading to Death by System |
| | | Organ Class and Preferred Term (Safety Population) |
| 14.3.4 | | Laboratory |
| | 14.3.4.1 | Shift from Baseline in Hematology Results by Test and Visit |
| | | (Safety Population) |
| | 14.3.4.2 | Shift from Baseline in Chemistry Results by Test and Visit (Safety |
| | | Population) |
| | 14.3.4.3 | Observed and Change from Baseline in Vital Sign Results by Test |
| | | and Visit (Safety Population) |
| | 14.3.4.4.1 | Shift from Baseline in 12-Lead ECG Overall Interpretation by Visit |
| | | (Safety Population) |
| | 14.3.4.4.2 | Summary of QTcF Interval (msec) by Visit and Result Category |
| | | (Safety Population) |

# **List of Figures**

| ICH | Figure | |
|---|---|---|
| Heading | Number | Figure Description |
| 14.3.4 | | Figure Description Laboratory Line Plots of Mean (+/- SD) Hematology Results vs. Time by Test (Safety Population) Line Plots of Mean (+/- SD) Chemistry Results vs. Time by Test (Safety Population) Line Plots of Mean (+/- SD) Vital Sign Results vs. Time by Test (Safety Population) Line Plots of Mean (+/- SD) 12-Lead ECG Results vs. Time by |
| | 14.3.4.1 | Line Plots of Mean (+/- SD) Hematology Results vs. Time by Test |
| | | Inber Figure Description Laboratory 3.4.1 Line Plots of Mean (+/- SD) Hematology Results vs. Time by Test (Safety Population) 3.4.2 Line Plots of Mean (+/- SD) Chemistry Results vs. Time by Test (Safety Population) 3.4.3 Line Plots of Mean (+/- SD) Vital Sign Results vs. Time by Test (Safety Population) |
| | 14.3.4.2 | Line Plots of Mean (+/- SD) Chemistry Results vs. Time by Test |
| | | (Safety Population) |
| | 14.3.4.3 | Line Plots of Mean (+/- SD) Vital Sign Results vs. Time by Test |
| | | (Safety Population) |
| | 14.3.4.4 | Line Plots of Mean (+/- SD) 12-Lead ECG Results vs. Time by |
| | | Test (Safety Population) |

# **List of Data Listings**

| ICH Heading | Listing | |
|-------------|----------|-------------------------------------------------|
| | Number | Listing Description |
| 16.2 | | SUBJECT DATA LISTINGS |
| 16.2.1 | | Discontinued Subjects |
| | 16.2.1 | Subject Disposition |
| 16.2.2 | | Protocol Deviations |
| | 16.2.2 | Protocol Deviations |
| 16.2.3 | | Subjects Excluded from the Safety Analysis |
| | 16.2.3 | Inclusion/Exclusion Criteria |
| 16.2.4 | | Demographic and Baseline Data |
| | 16.2.4.1 | Demographic and Baseline Characteristics |
| | 16.2.4.2 | Medical History |
| | 16.2.4.3 | Prior and Concomitant Medications |
| 16.2.5 | | Compliance and/or Drug Concentration Data |
| | 16.2.5.1 | Exposure and Treatment Compliance |
| | 16.2.5.2 | Treatment Diary |
| | 16.2.5.3 | Plasma Collection for Measurement of Quinine |
| 16.2.6 | | Individual Efficacy Response Data |
| | 16.2.6.1 | PCR Results |
| | 16.2.6.2 | Symptom Scores |
| | 16.2.6.3 | Seroconversion |
| 16.2.7 | | Adverse Events listings |
| | 16.2.7.1 | Adverse Events |
| | 16.2.7.2 | Serious Adverse Events |
| | 16.2.7.3 | Adverse Events Leading to Study Discontinuation |
| | 16.2.7.4 | Deaths |
| 16.2.8 | | Laboratory and Other Data |
| | 16.2.8.1 | Hematology |
| | 16.2.8.2 | Chemistry |
| | 16.2.8.3 | Vital Signs |
| | 16.2.8.4 | 12-Lead Electrocardiogram |
| | 16.2.8.5 | Physical Examination |
| | 16.2.8.6 | Pregnancy Test |



#### Table 14.1.1.1 Subject Disposition (All Subjects)

| tudy Site<br>Subject Status | GLS-1200 | Placebo | Overall |
|-----------------------------|-----------|-----------|-----------|
| verall | | | |
| creened | | | xx |
| creen Failures | | | XX |
| T Population [1] | XX | xx | XX |
| afety Population [2] | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| P Population [3] | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| ompleted the study [4] | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| iscontinued the study | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Reason for discontinuation | | | |
| <reason #1=""></reason> | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <reason #2=""></reason> | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <reason #3=""></reason> | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| te 101 | | | |
| te 108 | | | |

Percentages are based on the ITT Population.

- [1] The Intent-to-treat (ITT) Population includes all randomized to treatment allocation.
- [2] The Safety Population includes all subjects who received at least one dose of study treatment.
- [3] The Per-protocol (PP) Population includes all subjects who completed the trial, received >=90% of the study treatments, and have no significant protocol deviations. Trial completion is defined as either completing Week 4 or meeting the study endpoint of PCR confirmed SARS-CoV-2 infection.
- [4] Study completion is defined as completing all visits regardless of drug compliance.

Reference: Listing 16.2.1

Programming note: Sort discontinuation reasons by descending overall frequency. List all reasons per CRF page.

Table 14.1.1.2 Reason for Screen Failure (All Screen Failure Subjects)

| Study Site Reason | Overall |
|-------------------------|-----------|
| | (xx) |
| Overall | |
| <reason #1=""></reason> | x (xx.x%) |
| <reason #2=""></reason> | x (xx.x%) |
| <reason #3=""></reason> | x (xx.x%) |
| Site 101 | |
| <reason #1=""></reason> | x (xx.x%) |
| :Reason #2> | x (xx.x%) |
| Reason #3> | x (xx.x%) |
| Site 108 | |
| <reason #1=""></reason> | x (xx.x%) |
| <reason #2=""></reason> | x (xx.x%) |
| <reason #3=""></reason> | x (xx.x%) |

Reference: Listing 16.2.3 and Listing 16.2.1

Programming note: Sort screen failure reasons by descending overall frequency. List all reasons per CRF page.

Table 14.1.2 Demographic and Baseline Characteristics (Safety Population)

| Study Site | GLS-1200 | Placebo | Overall |
|---|---|---|---|
| Characteristic | (N=XX) | (N=XX) | (N=XX) |
| Overall | | | |
| Age (years) | | | |
| n | XX | xx | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | xx.x | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| <65 years | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| >=65 years | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Sex | | | |
| Male | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Female | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Race | | | |
| American Indian or Alaskan Native | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Asian | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Black or African American | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Native Hawaiian or Other Pacific Islander | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| White | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Other | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Ethnicity | | | |
| Hispanic or Latino | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| Not Hispanic or Latino | x (xx.x%) | x (xx.x%) | x (xx.x%) |

Baseline is the last non-missing value prior to first dose of study treatment. Reference: Listing 16.2.4.1 and Listing 16.2.1

date time

Table 14.1.2

Demographic and Baseline Characteristics
(Safety Population)

| paracteristic | GLS-1200 | Placebo | Overall |
|---------------|-------------|-------------|-------------|
| | (N=XX) | (N=XX) | (N=XX) |
| eight (cm) | | | |
| n | XX | xx | XX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | XX.X | xx.x | XX.X |
| Min, Max | xx, xx | XX, XX | xx, xx |
| eight (kg) | | | |
| n | XX | xx | XX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | XX.X | xx.x | XX.X |
| Min, Max | xx, xx | xx, xx | xx, xx |
| ЛI (kg/m^2) | | | |
| n | XX | xx | XX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | XX.X | xx.x | XX.X |
| Min, Max | xx, xx | XX, XX | xx, xx |
| re 101 | | | |
| ne 108 | | | |

Baseline is the last non-missing value prior to first dose of study treatment. Reference: Listing 16.2.4.1 and Listing 16.2.1

date

time

Table 14.1.3 Medical History (Safety Population)

| udy Site | GLS-1200 | | Overall |
|------------------------------------------|-----------|-----------|-----------|
| | (N=XX) | (N=XX) | (N=XX) |
| stem Organ Class | | | |
| Preferred Term | | | |
| verall | | | |
| bjects with at least one medical history | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| ystem Organ Class #1> | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #1="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| ystem Organ Class #2> | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #1="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) |

Site 101

.

.

Site 108

MedDRA = Medical Dictionary for Regulatory Activities; SOC = System Organ Class; PT = Preferred Term.

Medical history terms are coded using MedDRA version 23.0 and ordered by descending order of overall incidence of SOC and overall incidence of PT within each SOC. At each level of summation (overall, SOC, PT), subjects reporting more than one medical history term are counted only once.

Reference: Listing 16.2.4.2 and Listing 16.2.1

date

time

#### Table 14.1.4 Concomitant Medications (Safety Population)

| Study Site | GLS-1200 | Placebo |
|---------------------------------------|-----------|-----------|
| 470.0 | (N=XX) | (N=XX) |
| ATC Class | | |
| Preferred Name | | |
| Overall | | |
| Subjects who received any concomitant | | |
| medications | x (xx.x%) | x (xx.x%) |
| <atc #="" 1="" class=""></atc> | x (xx.x%) | x (xx.x%) |
| <preferred #1="" name=""></preferred> | x (xx.x%) | x (xx.x%) |
| <preferred #2="" name=""></preferred> | x (xx.x%) | x (xx.x%) |
| <preferred #3="" name=""></preferred> | x (xx.x%) | x (xx.x%) |
| <atc #="" 2="" class=""></atc> | x (xx.x%) | x (xx.x%) |
| <preferred #1="" name=""></preferred> | x (xx.x%) | x (xx.x%) |
| <preferred #2="" name=""></preferred> | x (xx.x%) | x (xx.x%) |
| <preferred #3="" name=""></preferred> | x (xx.x%) | x (xx.x%) |
| • | | |
| Site 101 | | |
| Site 108 | | |
| • | | |
| · | | |

A concomitant medication is any medication that was ongoing or started on or after the date of first dose.

Medications are coded using WHODrug Global (March 2020) and ordered by descending order of overall incidence of ATC class and overall incidence of preferred name within each class. At each level of summation (overall, ATC class, preferred name), subjects reporting more than one medication are counted only once.

Reference: Listing 16.2.4.3 and Listing 16.2.1

date time

Programming Note: Sort table by descending overall count of ATC class and descending overall count of preferred name within each class.

#### Table 14.1.5 **Exposure and Treatment Compliance** (Safety Population)

| | GLS-1200 | Placebo |
|--------------------------------|--------------|--------------|
| | (N=XX) | (N=XX) |
| erall | | |
| uration of exposure (days) [1] | | |
| n | XX | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | xx.x |
| Min, Max | xx, xx | xx, xx |
| otal number of doses taken | | |
| n | XX | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx |
| atal number of doses missed | | |
| n | XX | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX |
| eatment compliance [2] | | |
| n | XX | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X |
| Min, Max | xx, xx | XX, XX |
| <50% | x (xx.x%) | x (xx.x%) |
| 50%-80% | x (xx.x%) | x (xx.x%) |
| >80% | x (xx.x%) | x (xx.x%) |
| re 101 | | |
| e 108 | | |

<sup>[1]</sup> Duration of exposure is defined as the date of last dose minus the date of first dose + 1.
[2] Treatment compliance is defined as the total number of doses taken divided by the total number of planned doses times 100. Reference: Listing 16.2.5.1 and Listing 16.2.1

Table 14.2.1.1 Incidence of SARS-CoV-2 Infection by Visit (ITT Population)

| | GLS-1200 | Placebo<br>(N=XX) | p-value [1] |
|---|---|---|---|
| | (N=XX) | | |
| reatment Success [2] | x (xx.x%) | x (xx.x%) | X.XXX |
| reatment Failure [3] | x (xx.x%) | x (xx.x%) | |
| Lost to follow-up | x (xx.x%) | x (xx.x%) | |
| Required recue therapy | x (xx.x%) | x (xx.x%) | |
| Discontinued study prior to completion of Week 4 | x (xx.x%) | x (xx.x%) | |
| Tested positive for SARS-CoV-2 infection at any time up to Week 4 | x (xx.x%) | x (xx.x%) | |
| Had missing PCR result at any visit up to Week 4 | x (xx.x%) | x (xx.x%) | |
| Died | x (xx.x%) | x (xx.x%) | |
| Neek 0 PCR Result | | | |
| n | Х | x | |
| Negative | x (xx.x%) | x (xx.x%) | |
| Positive | x (xx.x%) | x (xx.x%) | |
| Missing | x (xx.x%) | x (xx.x%) | |
| Week 2 PCR Result | | | |
| n | Х | x | |
| Negative | x (xx.x%) | x (xx.x%) | |
| Positive | x (xx.x%) | x (xx.x%) | |
| Missing | x (xx.x%) | x (xx.x%) | |

<sup>[1]</sup> The p-value is calculated using a Fisher's exact test.

Programming note: Continue for remaining visits. Repeat for Table 14.2.1.2 Incidence of SARS-CoV-2 Infection (PP Population).

<sup>[2]</sup> Subjects who test negative for SARS-CoV-2 infection at Weeks 2 and 4 are considered treatment successes.

<sup>[3]</sup> Subjects who met any of the reasons listed are considered treatment failures. Subjects who fail treatment for multiple reasons are counted once for each reason. Reference: Listing 16.2.6.1

Table 14.2.2
Incidence of Individual Symptoms and Average Number of Days with Symptoms by Visit Interval (ITT Population)

| ymptom | GLS-1200 | Placebo |
|---|---|---|
| | (N=XX) | (N=XX) |
| ubjects who reported Body Aches at least once from Day 1 to Week 2 | x (xx.x%) | x (xx.x%) |
| ubjects who reported Body Aches at least once from Week 2 to Week 4 | x (xx.x%) | x (xx.x%) |
| ubjects who reported Body Aches at least once from Week 4 to Week 6 | x (xx.x%) | x (xx.x%) |
| bjects who reported Body Aches at least once during the overall treatment phase [1] | x (xx.x%) | x (xx.x%) |
| umber of days subjects reported Body Aches from Day 1 to Week 2 | | |
| n | X | х |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx |
| umber of days subjects reported Body Aches from Week 2 to Week 4 | | |
| n | Х | х |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx |
| umber of days subjects reported Body Aches from Week 4 to Week 6 | | |
| n | Х | X |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X |
| Min, Max | xx, xx | xx, xx |
| umber of days subjects reported Body Aches during the overall treatment phase [1] | | |
| n | x | х |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X |
| Min, Max | xx, xx | xx, xx |

Percentages are based on the ITT Population.

Number of days summaries include subjects who experienced no symptoms, reported as 0 days.

[1] Includes the time from Day 1 to Week 4.

Reference: Listing 16.2.6.2.1

Programming Note: Continue for each individual symptom.

#### Table 14.2.3 Cumulative Incidence of SARS-CoV-2 Seroconversion by Visit (ITT Population)

| sit | GLS-1200 | Placebo |
|---------------|-----------|-----------|
| Seroconverted | (N=XX) | (N=XX) |
| reek 2 | | |
| n | х | x |
| Yes | x (xx.x%) | x (xx.x%) |
| No | x (xx.x%) | x (xx.x%) |
| eek 4 | | |
| n | Х | х |
| Yes | x (xx.x%) | x (xx.x%) |
| No | x (xx.x%) | x (xx.x%) |
| reek 6 | | |
| n | Х | Х |
| Yes | x (xx.x%) | x (xx.x%) |
| No | x (xx.x%) | x (xx.x%) |

The incidence of seroconversion is summarized based on results obtained at or prior to the visit.

Reference: Listing 16.2.6.3

#### Table 14.3.1.1 Overall Summary of Adverse Events (Safety Population)

| | GLS-1200 | Placebo |
|---|---|---|
| | (N=XX) | (N=XX) |
| | n (%) [95% Cl] | n (%) [95% CI] |
| ubjects with any TEAE | x (xx.x%) [xx.x% - xx.x%] | x (xx.x%) [xx.x% - xx.x%] |
| ubjects whose strongest TEAE relationship to study drug is related [1] | x (xx.x%) [xx.x% - xx.x%] | x (xx.x%) [xx.x% - xx.x%] |
| ubjects whose strongest TEAE relationship to study drug is not related [2] | x (xx.x%) [xx.x% - xx.x%] | x (xx.x%) [xx.x% - xx.x%] |
| ubjects whose maximum TEAE severity grade is Mild [3] | x (xx.x%) [xx.x% - xx.x%] | x (xx.x%) [xx.x% - xx.x%] |
| ubjects whose maximum TEAE severity grade is Moderate [3] | x (xx.x%) [xx.x% - xx.x%] | x (xx.x%) [xx.x% - xx.x%] |
| ubjects whose maximum TEAE severity grade is Severe [3] | x (xx.x%) [xx.x% - xx.x%] | x (xx.x%) [xx.x% - xx.x%] |
| ibjects with any SAE | x (xx.x%) [xx.x% - xx.x%] | x (xx.x%) [xx.x% - xx.x%] |
| ubjects with any serious TEAE | x (xx.x%) [xx.x% - xx.x%] | x (xx.x%) [xx.x% - xx.x%] |
| ubjects with any TEAE leading to study discontinuation | x (xx.x%) [xx.x% - xx.x%] | x (xx.x%) [xx.x% - xx.x%] |
| ubjects with any TEAE leading to death | x (xx.x%) [xx.x% - xx.x%] | x (xx.x%) [xx.x% - xx.x%] |

AE = adverse event; SAE = Serious Adverse Event; TEAE = Treatment-Emergent Adverse Event; CI = Confidence Interval

The 95% CIs for the subject percentages are calculated using an exact binomial distribution.

[1] Related TEAEs are those with a relationship of related, possibly related, or probably related. If the relationship is missing, it is considered related.

time

[2] Not related TEAEs are those with a relationship of unlikely related or not related.

[3] Severity grades are determined according to the NCI Common Terminology Criteria for Adverse Events version 5.0.

Reference: Listing 16.2.7.1

Table 14.3.1.2

Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population)

| ystem Organ Class | GLS-1200 | Placebo |
|---------------------------------------|-----------|-----------|
| Preferred Term | (N=XX) | (N=XX) |
| ubjects with at least one TEAE | x (xx.x%) | x (xx.x%) |
| System Organ Class #1> | x (xx.x%) | x (xx.x%) |
| <preferred #1="" term=""></preferred> | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) |
| System Organ Class #2> | x (xx.x%) | x (xx.x%) |
| <preferred #1="" term=""></preferred> | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) |

AE=adverse event; TEAE = Treatment-Emergent Adverse Event; MedDRA = Medical Dictionary for Regulatory Activities.

AEs are coded using MedDRA version 23.0 and ordered by descending order of overall incidence of SOC and overall incidence of PT within each SOC. At each level of summation (overall, SOC, PT), subjects reporting more than one TEAE are counted only once.

Reference: Listing 16.2.7.1

Table 14.3.1.3

Treatment-Emergent Adverse Events by System Organ Class, Preferred Term, and Strongest Relationship to Study Drug (Safety Population)

| System Organ Class Preferred Term | GLS | 5-1200 | Pla | acebo |
|---|---|---|---|---|
| | (N=XX) | | (N=XX) | |
| | Related | Not Related | Related | Not Related |
| Subjects with at least one TEAE | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <system #1="" class="" organ=""></system> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #1="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <system #2="" class="" organ=""></system> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #1="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |

AE=adverse event; TEAE = Treatment-Emergent Adverse Event; MedDRA = Medical Dictionary for Regulatory Activities.

AEs are coded using MedDRA version 23.0 and ordered by descending order of overall incidence of SOC and overall incidence of PT within each SOC. At each level of summation (overall, SOC, PT), subjects reporting more than one TEAE are counted only once using the strongest relationship.

Related TEAEs are those with a relationship of related, possibly related, or probably related. If the relationship is missing, it is considered related. Not Related TEAEs are those with a relationship of unlikely related or not related.

Reference: Listing 16.2.7.1

date

time
GeneOne Life Science Inc.
Protocol: T2R-002

Table 14.3.1.4

Treatment-Emergent Adverse Events by System Organ Class, Preferred Term, and Maximum Severity Grade (Safety Population)

| System Organ Class | | GLS-1200 | | | Placebo | |
|---|---|---|---|---|---|---|
| Preferred Term | | (N=XX) | | | (N=XX) | |
| | Mild | Moderate | Severe | Mild | Moderate | Severe |
| Subjects with at least one TEAE | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <system #1="" class="" organ=""></system> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #1="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| System Organ Class #2> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #1="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) | x (xx.x%) |

AE=adverse event; TEAE = Treatment-Emergent Adverse Event; MedDRA = Medical Dictionary for Regulatory Activities

AEs are coded using MedDRA version 23.0 and ordered by descending order of overall incidence of SOC and overall incidence of PT within each SOC. At each level of summation (overall, SOC, PT), subjects reporting more than one TEAE are counted only once using the highest grade.

 $Severity\ grades\ are\ determined\ according\ to\ the\ NCI\ Common\ Terminology\ Criteria\ for\ Adverse\ Events\ version\ 5.0.$ 

Reference: Listing 16.2.7.1

Repeat Table 14.3.1.4 layout for:

Table 14.3.1.5

Related Treatment-Emergent Adverse Events by System Organ Class, Preferred Term, and Maximum Severity Grade (Safety Population)

Table 14.3.2.1 Serious Adverse Events by System Organ Class and Preferred Term (Safety Population)

| System Organ Class | GLS-1200 | Placebo |
|-------------------------------------------|-----------|-----------|
| Preferred Term | (N=XX) | (N=XX) |
| Subjects with at least one SAE | x (xx.x%) | x (xx.x%) |
| <system #1="" class="" organ=""></system> | x (xx.x%) | x (xx.x%) |
| <preferred #1="" term=""></preferred> | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) |
| System Organ Class #2> | x (xx.x%) | x (xx.x%) |
| <preferred #1="" term=""></preferred> | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) |

SAE=serious adverse event; MedDRA = Medical Dictionary for Regulatory Activities.

AEs are coded using MedDRA version 23.0 and ordered by descending order of overall incidence of SOC and overall incidence of PT within each SOC. At each level of summation (overall, SOC, PT), subjects reporting more than one AE are counted only once.

Reference: Listing 16.2.7.2

Table 14.3.2.2
Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population)

| system Organ Class | GLS-1200 | Placebo |
|----------------------------------------|-----------|-----------|
| Preferred Term | (N=XX) | (N=XX) |
| ubjects with at least one serious TEAE | x (xx.x%) | x (xx.x%) |
| System Organ Class #1> | x (xx.x%) | x (xx.x%) |
| <preferred #1="" term=""></preferred> | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) |
| System Organ Class #2> | x (xx.x%) | x (xx.x%) |
| <preferred #1="" term=""></preferred> | x (xx.x%) | x (xx.x%) |
| <preferred #2="" term=""></preferred> | x (xx.x%) | x (xx.x%) |

AE=adverse event; TEAE = Treatment-Emergent Adverse Event; MedDRA = Medical Dictionary for Regulatory Activities.

AEs are coded using MedDRA version 23.0 and ordered by descending order of overall incidence of SOC and overall incidence of PT within each SOC. At each level of summation (overall, SOC, PT), subjects reporting more than one TEAE are counted only once.

Reference: Listing 16.2.7.2

Table 14.3.2.3

Treatment-Emergent Adverse Events Leading to Study Discontinuation by System Organ Class and Preferred Term (Safety Population)

| GLS-1200 | Placebo |
|---|---|
| (N=XX) | (N=XX) |
| x (xx.x%) | x (xx.x%) |
| x (xx.x%) | x (xx.x%) |
| x (xx.x%) | x (xx.x%) |
| x (xx.x%) | x (xx.x%) |
| x (xx.x%) | x (xx.x%) |
| x (xx.x%) | x (xx.x%) |
| x (xx.x%) | x (xx.x%) |
| | (N=XX) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) x (xx.x%) |

AE=adverse event; TEAE = Treatment-Emergent Adverse Event; MedDRA = Medical Dictionary for Regulatory Activities

AEs are coded using MedDRA version 23.0 and ordered by descending order of overall incidence of SOC and overall incidence of PT within each SOC. At each level of summation (overall, SOC, PT), subjects reporting more than one TEAE are counted only once.

Reference: Listing 16.2.7.3

Table 14.3.2.4

Treatment-Emergent Adverse Events Leading to Death by System Organ Class and Preferred Term (Safety Population)

| (N=XX)<br>x (xx.x%)<br>x (xx.x%) | (N=XX)<br>x (xx.x%) |
|----------------------------------|------------------------|
| | , , |
| v (vv v%) | |
| Λ (ΛΛ·Λ/0) | x (xx.x%) |
| x (xx.x%) | x (xx.x%) |
| x (xx.x%) | x (xx.x%) |
| x (xx.x%) | x (xx.x%) |
| x (xx.x%) | x (xx.x%) |
| x (xx.x%) | x (xx.x%) |
| | x (xx.x%)<br>x (xx.x%) |

AE=adverse event; TEAE = Treatment-Emergent Adverse Event; MedDRA = Medical Dictionary for Regulatory Activities

AEs are coded using MedDRA version 23.0 and ordered by descending order of overall incidence of SOC and overall incidence of PT within each SOC. At each level of summation (overall, SOC, PT), subjects reporting more than one TEAE are counted only once.

Reference: Listing 16.2.7.4

Table 14.3.4.1 Shift from Baseline in Hematology Results by Test and Visit (Safety Population)

| est | | GLS-1200 | | | Placebo | |
|---|---|---|---|---|---|---|
| Visit | | (N=XX) | | | (N=XX) | |
| | | Baseline | | Baseline | | |
| | Low | Normal | High | Low | Normal | High |
| Test #1> (units) | | | | | | |
| Week 4 | | | | | | |
| n | | X | | | x | |
| Low | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Normal | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| High | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Baseline is the last non-missing value prior to first dose of study treatment.

Percentages are based on n, the number of subjects with both a baseline and post-baseline result at the visit.

Shifts are based on local labs from each site.

Reference: Listing 16.2.8.1

date

time

Programming Note: Continue for all hematology tests.

Repeat Table 14.3.4.1 layout for:

Table 14.3.4.2 Shift from Baseline in Chemistry Results by Test and Visit (Safety Population)

Table 14.3.4.3

Observed and Change from Baseline in Vital Sign Results by Test and Visit (Safety Population)

| Test | | GLS-1200 | | Placebo |
|---|---|---|---|---|
| Visit | | (N=XX) | | (N=XX) |
| | Observed | Change from Baseline | Observed | Change from Baseline |
| Test #1> (units) | | | | |
| Baseline | | | | |
| n | Х | | x | |
| Mean (SD) | xx.xx (xx.xxx) | | xx.xx (xx.xxx) | |
| Median | x.xx | | x.xx | |
| Min, Max | xx.x, xx.x | | xx.x, xx.x | |
| Week 2 | | | | |
| n | х | X | x | x |
| Mean (SD) | xx.xx (xx.xxx) | xx.xx (xx.xxx) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| Median | x.xx | x.xx | x.xx | x.xx |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | XX.X, XX.X |
| Week 4 | | | | |
| n | х | X | x | x |
| Mean (SD) | xx.xx (xx.xxx) | xx.xx (xx.xxx) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| Median | x.xx | x.xx | x.xx | x.xx |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | XX.X, XX.X |
| Week 6 | | | | |
| n | х | X | x | x |
| Mean (SD) | xx.xx (xx.xxx) | xx.xx (xx.xxx) | xx.xx (xx.xxx) | xx.xx (xx.xxx) |
| Median | x.xx | x.xx | x.xx | x.xx |
| Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |

Baseline is the last non-missing value prior to first dose of study treatment.

Reference: Listing 16.2.8.3

Programming Note: Continue for all vital sign tests.

#### Table 14.3.4.4.1 Shift from Baseline in 12-Lead ECG Overall Interpretation by Visit (Safety Population)

| | | GLS-1200 | | | Placebo | |
|---|---|---|---|---|---|---|
| | | (N=XX) | | | (N=XX) | |
| | | Baseline | | | Baseline | |
| | Normal | Abnormal NCS | Abnormal CS | Normal | Abnormal NCS | Abnormal CS |
| Veek 4 | | | | | | |
| n | | X | | | X | |
| Normal | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal NCS | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Abnormal CS | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

(N)CS = (Not) Clinically Significant.

Baseline is the last non-missing value prior to first dose of study treatment.

Percentages are based on n, the number of subjects with both a baseline and post-baseline result at the visit.

Reference: Listing 16.2.8.4

#### Table 14.3.4.4.2 Summary of QTcF Interval (msec) by Visit and Result Category (Safety Population)

| Visit<br>Result Category | GLS-1200<br>(N=XX) | Placebo<br>(N=XX) |
|---|---|---|
| Baseline | | |
| n | X | X |
| <=450 msec (males) or <=470 msec (females) | xx (xx.x) | xx (xx.x) |
| >450 msec (males) or >470 msec (females) | xx (xx.x) | xx (xx.x) |
| Week 4 | | |
| n | X | X |
| <=450 msec (males) or <=470 msec (females) | xx (xx.x) | xx (xx.x) |
| >450 msec (males) or >470 msec (females) | xx (xx.x) | xx (xx.x) |
| Change from baseline <=60 msec | xx (xx.x) | xx (xx.x) |
| Change from baseline >60 msec | xx (xx.x) | xx (xx.x) |

Baseline is the last non-missing value prior to first dose of study treatment.

Percentages are based on n, the number of subjects with a baseline and post-baseline (for Week 4) result at the visit.

Reference: Listing 16.2.8.4



Figure 14.3.4.1 Line Plots of Mean (+/-SD) Hematology Results vs. Time by Test (Safety Population)



Reference: Listing 16.2.8.1

Programming Note: Display each hematology test on a separate page. Repeat Figure 14.3.4.1 layout for: Line Plots of Mean (+/-SD) Chemistry Results vs. Time by Test Safety Population

Figure 14.3.4.3 Line Plots of Mean (+/-SD) Vital Sign Results vs. Time by Test Safety Population

Figure 14.3.4.4 Line Plots of Mean (+/-SD) 12-Lead ECG Results vs. Time by Test Safety Population



Listing 16.2.1 Subject Disposition

Treatment: GLS-1200, Placebo

| Subject ID | Study Site | Informed<br>Consent<br>Date | Randomization<br>Date | ITT<br>Population [1] | Safety<br>Population [2] | PP<br>Population [3] | First Dose<br>Date | Study<br>Completion<br>Status | Study Completion or<br>Discontinuation<br>Date<br>(Study Day) |
|---|---|---|---|---|---|---|---|---|---|
| xxxxx | xxxxx | yyyy-mm-dd | yyyy-mm-dd | Yes/No | Yes/No | Yes/No | yyyy-mm-dd | xxxxxxxxx | yyyy-mm-dd (xx) |
| xxxxx | xxxxx | yyyy-mm-dd | yyyy-mm-dd | Yes/No | Yes/No | Yes/No | yyyy-mm-dd | | yyyy-mm-dd (xx) |
| XXXXX | xxxxx | yyyy-mm-dd | yyyy-mm-dd | Yes/No | Yes/No | Yes/No | yyyy-mm-dd | xxxxxxxxx | yyyy-mm-dd (xx) |
| XXXXX | xxxxx | yyyy-mm-dd | yyyy-mm-dd | Yes/No | Yes/No | Yes/No | yyyy-mm-dd | xxxxxxxxx | yyyy-mm-dd (xx) |
| xxxxx | xxxxx | yyyy-mm-dd | yyyy-mm-dd | Yes/No | Yes/No | Yes/No | yyyy-mm-dd | xxxxxxxxx | yyyy-mm-dd (xx) |
| xxxxx | xxxxx | yyyy-mm-dd | yyyy-mm-dd | Yes/No | Yes/No | Yes/No | yyyy-mm-dd | xxxxxxxxx | yyyy-mm-dd (xx) |
| xxxxx | XXXXX | yyyy-mm-dd | yyyy-mm-dd | Yes/No | Yes/No | Yes/No | yyyy-mm-dd | xxxxxxxxx | yyyy-mm-dd (xx) |
| xxxxx | XXXXX | yyyy-mm-dd | yyyy-mm-dd | Yes/No | Yes/No | Yes/No | yyyy-mm-dd | xxxxxxxxx | yyyy-mm-dd (xx) |

<sup>[1]</sup> The Intent-to-treat (ITT) Population includes all randomized to treatment allocation.

date time

<sup>[2]</sup> The Safety Population includes all subjects who received at least one dose of study treatment.

<sup>[3]</sup> The Per-protocol (PP) Population includes all subjects who completed the trial, received >=90% of the study treatments, and have no significant protocol deviations. Trial completion is defined as either completing Week 4 or meeting the study endpoint of PCR confirmed SARS-CoV-2 infection.

Listing 16.2.2 Protocol Deviations

Treatment: GLS-1200, Placebo

| Subject ID | Deviation Date<br>(Study Day) | Deviation Category | Description |
|---|---|---|---|
| | (Study Day) | | |
| xxxxx | yyyy-mm-dd (xx) | Major/Minor | XXXXXX |
| XXXXX | yyyy-mm-dd (xx) | Major/Minor | XXXXXX |
| XXXXX | yyyy-mm-dd (xx) | Major/Minor | xxxxxx |
| XXXXX | yyyy-mm-dd (xx) | Major/Minor | XXXXXX |
| XXXXX | yyyy-mm-dd (xx) | Major/Minor | xxxxxx |
| XXXXX | yyyy-mm-dd (xx) | Major/Minor | XXXXXX |
| XXXXX | yyyy-mm-dd (xx) | Major/Minor | xxxxxx |
| (XXXXX | yyyy-mm-dd (xx) | Major/Minor | XXXXXX |

Listing 16.2.3 Inclusion/Exclusion Criteria

Treatment: GLS-1200, Placebo

| Subject ID | All eligibility criteria met | Criterion not met | Criterion Description |
|---|---|---|---|
| | v. 60 | | |
| xxxxxx | Yes/No | Inclusion xx/Exclusion xx | XXXXXXXX |
| XXXXXX | Yes/No | Inclusion xx/Exclusion xx | XXXXXXXX |
| XXXXXX | Yes/No | Inclusion xx/Exclusion xx | XXXXXXX |
| XXXXXX | Yes/No | Inclusion xx/Exclusion xx | xxxxxxx |
| XXXXXX | Yes/No | Inclusion xx/Exclusion xx | xxxxxxx |
| xxxxxx | Yes/No | Inclusion xx/Exclusion xx | xxxxxxx |
| xxxxxx | Yes/No | Inclusion xx/Exclusion xx | xxxxxxx |
| xxxxxx | Yes/No | Inclusion xx/Exclusion xx | xxxxxxx |
| Source: \\xx\xxx\xxx\xxx\xxx | xxxx\xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | time | |

Programming Note: If more than one criterion ID is selected for a subject, list each one on a separate line.

### Protocol: T2R-002

## Listing 16.2.4.1 Demographic and Baseline Characteristics

Treatment: GLS-1200, Placebo

| Subject ID | Age | Sex | Race | Ethnicity | Height | Weight | BMI |
|---|---|---|---|---|---|---|---|
| | (years) | | | | (cm) | (kg) | (kg/m^2) |
| xxxxxx | XX | Male/Female | xxxxxxxxxxx | xxxxxxxxxx | xx.x | xx.x | xx.x |
| XXXXXX | xx | Male/Female | XXXXXXXXXXX | xxxxxxxxxxx | XX.X | XX.X | XX.X |
| XXXXXX | xx | Male/Female | XXXXXXXXXXX | XXXXXXXXXXX | xx.x | xx.x | XX.X |
| xxxxxx | XX | Male/Female | XXXXXXXXXXX | XXXXXXXXXXX | XX.X | XX.X | XX.X |
| XXXXXX | XX | Male/Female | XXXXXXXXXXX | XXXXXXXXXXX | XX.X | XX.X | XX.X |
| XXXXXX | XX | Male/Female | XXXXXXXXXXX | XXXXXXXXXXX | XX.X | XX.X | XX.X |
| 100000 | vo. | Male/Female | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | VV V | VIV. V | VII. V |
| XXXXXX | XX | • | xxxxxxxxxxx | xxxxxxxxxxx | XX.X | xx.x | XX.X |
| XXXXXX | XX | Male/Female | XXXXXXXXXXX | XXXXXXXXXXX | XX.X | XX.X | XX.X |

Baseline is the last non-missing value prior to first dose of study treatment.

date time

Listing 16.2.4.2 Medical History

Treatment: GLS-1200, Placebo

| Subject ID | Any medical history | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Start Date | Ongoing | Stop Date |
|---|---|---|---|---|---|
| xxxxxx | Yes/No | xxxxxxxxx/<br>xxxxxxxxx/<br>xxxxxxxxx | yyyy-mm-dd | Yes/No | yyyy-mm-dd |
| | | xxxxxxxxx/<br>xxxxxxxxx/<br>xxxxxxxxx | yyyy-mm-dd | Yes/No | yyyy-mm-dd |
| XXXXXX | Yes/No | xxxxxxxxx/<br>xxxxxxxxx/<br>xxxxxxxxx | yyyy-mm-dd | Yes/No | yyyy-mm-dd |
| | | xxxxxxxxxx/<br>xxxxxxxxxx/<br>xxxxxxxxx | yyyy-mm-dd | Yes/No | yyyy-mm-dd |
| xxxxxx | Yes/No | xxxxxxxxx/<br>xxxxxxxxx/<br>xxxxxxxxx | yyyy-mm-dd | Yes/No | yyyy-mm-dd |
| | | xxxxxxxxxx/<br>xxxxxxxxxx/<br>xxxxxxxxx | yyyy-mm-dd | Yes/No | yyyy-mm-dd |

MedDRA = Medical Dictionary for Regulatory Activities.
Medical history terms are coded using MedDRA version 23.0.

date

time

## Listing 16.2.4.3 Prior and Concomitant Medications

Treatment: GLS-1200, Placebo

| Subject ID | ATC Class/<br>Preferred Name/ | Start Date<br>(Study Day)/ | Dose | Units | Route | Frequency | Indication |
|---|---|---|---|---|---|---|---|
| | Verbatim Term | End Date | | | | | |
| | | (Study Day) | | | | | |
| xxxxxx | xxxxxxxxx/ | yyyy-mm-dd (xx)/ | xxxxxxxxx | xxxxxxxxx | XXXXXXXXX | XXXXXXXXX | XXXXXXXXX |
| | xxxxxxxxx/ | yyyy-mm-dd (xx) | | | | | |
| | xxxxxxxx | | | | | | |
| | xxxxxxxxxx/ | yyyy-mm-dd (xx)/ | xxxxxxxxx | XXXXXXXXX | XXXXXXXXX | XXXXXXXXX | xxxxxxxxx |
| | xxxxxxxxx/ | yyyy-mm-dd (xx) | | | | | |
| | XXXXXXXX | | | | | | |
| xxxxxx | xxxxxxxxxx/ | yyyy-mm-dd (xx)/ | xxxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxxx |
| | xxxxxxxxx/ | yyyy-mm-dd (xx) | | | | | |
| | xxxxxxxx* | 7777 | | | | | |
| | xxxxxxxxxx/ | yyyy-mm-dd (xx)/ | xxxxxxxxx | XXXXXXXXX | xxxxxxxxx | XXXXXXXXX | xxxxxxxxx |
| | xxxxxxxxx/ | yyyy-mm-dd (xx) | | | | | |
| | xxxxxxxx | ,,,, | | | | | |
| XXXXXX | xxxxxxxxxx/ | yyyy-mm-dd (xx)/ | xxxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxxx |
| ***** | xxxxxxxxx/ | yyyy-mm-dd (xx) | ****** | ********** | ********* | ********* | ****** |
| | xxxxxxxx | yyyy mm da (xx) | | | | | |
| | xxxxxxxxxx/ | yyyy-mm-dd (xx)/ | xxxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxxx |
| | xxxxxxxxx/ | yyyy-mm-dd (xx)/ | ΛΛΛΛΛΛΛΛΛ | ΛΛΛΛΛΛΛΛΛ | ΛΛΛΛΛΛΛΛΛ | ΛΛΛΛΛΛΛΛΛ | ΛΛΛΛΛΛΛΛΛ |
| | xxxxxxxx | yyyy | | | | | |

Medications are coded using WHODrug Global (March 2020).

Prior medications are denoted by \*.

A prior medication is defined as a medication that was administered up to 8 weeks prior to first dose of study treatment. A concomitant medication is any medication that is ongoing or started on or after the date of first dose.

time

## Listing 16.2.5.1 Exposure and Treatment Compliance

Treatment: GLS-1200, Placebo

| Subject ID | Date of first dose | Date of last dose | Duration of Exposure (days) [1] | Number of Days<br>with At Least One Dose Taken | Total Doses Taken | Total Doses<br>Missed | Treatment Compliance [2] |
|---|---|---|---|---|---|---|---|
| xxxxx | yyyy-mm-dd | yyyy-mm-dd | XX | XX | xx | XX | xx% |
| xxxxxx | yyyy-mm-dd | yyyy-mm-dd | XX | XX | xx | XX | xx% |
| xxxxxx | yyyy-mm-dd | yyyy-mm-dd | XX | XX | XX | XX | xx% |
| xxxxxx | yyyy-mm-dd | yyyy-mm-dd | XX | XX | XX | XX | xx% |
| (XXXXX | yyyy-mm-dd | yyyy-mm-dd | XX | XX | xx | XX | xx% |
| xxxxx | yyyy-mm-dd | yyyy-mm-dd | XX | XX | xx | XX | xx% |
| (XXXXX | yyyy-mm-dd | yyyy-mm-dd | XX | XX | xx | XX | xx% |
| xxxxx | yyyy-mm-dd | yyyy-mm-dd | XX | XX | XX | xx | xx% |
| | 1111 | 7777 | | | | | |

<sup>[1]</sup> Duration of exposure is defined as the date of last dose minus the date of first dose + 1.

date

time

<sup>[2]</sup> Treatment compliance is defined as the total number of doses taken divided by the total number of planned doses times 100.

Listing 16.2.5.2 Treatment Diary

Treatment: GLS-1200, Placebo

| Subject ID | Day | Date (Study Day) | Dose 1 Taken | Dose 2 Taken | Dose 3 Taken | Diary Comments | SARS-CoV-2 Exposures:<br># Suspected | SARS-CoV-2 Exposures: # Known |
|---|---|---|---|---|---|---|---|---|
| | | | | | | | · | |
| XXXXXX | xx | yyyy-mm-dd (xx) | Yes/No | Yes/No | Yes/No | xxxxxxx | XX | XX |
| | XX | yyyy-mm-dd (xx) | Yes/No | Yes/No | Yes/No | xxxxxxxx | xx | XX |
| | XX | yyyy-mm-dd (xx) | Yes/No | Yes/No | Yes/No | XXXXXXXX | xx | XX |
| | XX | yyyy-mm-dd (xx) | Yes/No | Yes/No | Yes/No | XXXXXXXX | xx | XX |
| | XX | yyyy-mm-dd (xx) | Yes/No | Yes/No | Yes/No | xxxxxxxx | xx | XX |
| | XX | yyyy-mm-dd (xx) | Yes/No | Yes/No | Yes/No | XXXXXXXX | xx | XX |
| | XX | yyyy-mm-dd (xx) | Yes/No | Yes/No | Yes/No | XXXXXXXX | xx | XX |
| | XX | yyyy-mm-dd (xx) | Yes/No | Yes/No | Yes/No | xxxxxxxx | xx | xx |

date time

Listing 16.2.5.3 Plasma Collection for Measurement of Quinine

Treatment: GLS-1200, Placebo

| Subject ID | Visit | Plasma Collected | Collection Date/Time<br>(Study Day) | Date of Last Spray<br>Administration<br>(Study Day) | Test Result<br>(unit) |
|---|---|---|---|---|---|
| xxxxx | Week 2 | Yes/No | yyyy-mm-dd hh:mm<br>(xx) | уууу-mm-dd<br>(xx) | xx.x |
| xxxxx | Week 2 | Yes/No | yyyy-mm-dd hh:mm<br>(xx) | уууу-mm-dd<br>(xx) | xx.x |
| xxxxxx | Week 2 | Yes/No | yyyy-mm-dd hh:mm<br>(xx) | уууу-mm-dd<br>(xx) | xx.x |
| xxxxx | Week 2 | Yes/No | yyyy-mm-dd hh:mm<br>(xx) | уууу-mm-dd<br>(xx) | xx.x |

Protocol: T2R-002

Listing 16.2.6.1 PCR Results

Treatment: GLS-1200, Placebo

| Subject ID | Visit | Nasopharyngeal Swabs for Viral PCR<br>Collected | Collection Date<br>(Study Day) | Test Result |
|---|---|---|---|---|
| xxxxxx | Day 0 | Yes/No | yyyy-mm-dd<br>(xx) | Negative/Positive |
| | Week 2 | Yes/No | yyyy-mm-dd<br>(xx) | Negative/Positive |
| | Week 4 | Yes/No | yyyy-mm-dd<br>(xx) | Negative/Positive |
| | Week 6 | Yes/No | yyyy-mm-dd<br>(xx) | Negative/Positive |

date

time

Listing 16.2.6.2 Symptom Scores

Treatment: GLS-1200, Placebo

| Subject ID | Day | Date | Fever | Cough | Sore<br>Throat | Headache | Shortness<br>of<br>Breath | Body<br>Aches | Fatigue | GI<br>Issues | Runny<br>Nose | Sneezing | Loss<br>of<br>Smell | Loss<br>of<br>Taste | Red<br>Eyes |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | xx | yyyy-mm-dd | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 |
| | XX | yyyy-mm-dd | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 |
| | xx | yyyy-mm-dd | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 |

0=No, 1=Yes

time

date

Listing 16.2.6.3 Seroconversion

Treatment: GLS-1200, Placebo

| Subject<br>ID | Visit | Serum for Viral Antibodies<br>Collected | Collection Date<br>(Study Day) | Titer | Seroconversion |
|---|---|---|---|---|---|
| xxxxxx | Day 0 | Yes/No | yyyy-mm-dd<br>(xx) | xx | Yes/No |
| | Week 2 | Yes/No | yyyy-mm-dd<br>(xx) | xx | Yes/No |
| | Week 4 | Yes/No | yyyy-mm-dd<br>(xx) | xx | Yes/No |
| | Week 6 | Yes/No | yyyy-mm-dd<br>(xx) | xx | Yes/No |

date

time

> Listing 16.2.7.1 Adverse Events

Treatment: GLS-1200, Placebo

| Subject ID | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Start Date<br>(Study Day)/<br>End Date<br>(Study Day) | Severity | Relationship | Action Taken | Serious | Outcome | Study Discontinuation | Treatment Required |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxxxxxxxxxxx/<br>xxxxxxxxxxxxxxx/<br>xxxxxxx | yyyy-mm-dd (xx)/<br>yyyy-mm-dd (xx) | Grade x | xxxxxxxxx | xxxxxxxxxx | Yes/No | xxxxxxxxx | Yes/No | Yes/No |
| XXXXXX | xxxxxxxxxxxxxxx/<br>xxxxxxxxxxxxxxxx/<br>xxxxxx | yyyy-mm-dd (xx)/<br>yyyy-mm-dd (xx) | Grade x | xxxxxxxxx | xxxxxxxxx | Yes/No | xxxxxxxxx | Yes/No | Yes/No |
| xxxxxx | XXXXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXXXX/<br>XXXXXX | yyyy-mm-dd (xx)/<br>yyyy-mm-dd (xx) | Grade x | xxxxxxxxx | xxxxxxxxx | Yes/No | xxxxxxxxx | Yes/No | Yes/No |

Severity grades are determined according to the NCI Common Terminology Criteria for Adverse Events version 5.0.

date

time

Programming Note: Sort by Treatment, Subject ID, AE start date and end date.

Repeat Layout of Listing 16.2.7.1 for:

Listing 16.2.7.3 Adverse Events Leading to Study Discontinuation

## Protocol: T2R-002 Listing 16.2.7.2 Serious Adverse Events

Treatment: GLS-1200, Placebo

| Subject ID | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Start Date<br>(Study Day) | End Date<br>(Study Day) | Severity | Relationship | Action Taken | SAE Criteria | Outcome | Study Discontinuation | Treatment<br>Required |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxxxxxxxxxxx/<br>xxxxxxxxxxxxxxx/<br>xxxxxxx | yyyy-mm-dd (xx) | yyyy-mm-dd (xx) | Grade x | xxxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxxx | Yes/No | Yes/No |
| xxxxxx | xxxxxxxxxxxxxxx/<br>xxxxxxxxxxxxxxx/<br>xxxxxx | yyyy-mm-dd (xx) | yyyy-mm-dd (xx) | Grade x | xxxxxxxxx | xxxxxxxxx | xxxxxxxxx | xxxxxxxxx | Yes/No | Yes/No |
| xxxxxx | xxxxxxxxxxxxxx/<br>xxxxxxxxxxxxxx/<br>xxxxxxxx | yyyy-mm-dd (xx) | yyyy-mm-dd (xx) | Grade x | xxxxxxxxx | XXXXXXXXX | XXXXXXXXX | xxxxxxxxx | Yes/No | Yes/No |
| xxxxxx | xxxxxxxxxxxxxx/<br>xxxxxxxxxxxxxx/<br>xxxxxxxx | yyyy-mm-dd (xx) | yyyy-mm-dd (xx) | Grade x | XXXXXXXXX | XXXXXXXXX | xxxxxxxxx | xxxxxxxxx | Yes/No | Yes/No |

SAE = Serious Adverse Event

date

time

Programming Note: Sort by Treatment, Subject ID, AE start date and end date.


Protocol: T2R-002

Listing 16.2.7.4 Deaths

Treatment: GLS-1200, Placebo

| Subject ID | Death Date | If Death is Due to AE, |
|---|---|---|
| | (Study Day) | AE Term/ Start Date (Study Day) |
| XXXXXX | yyyy-mm-dd (xx) | xxxxxxxxxxxx/ yyyy-mm-dd (xx) |
| xxxxxx | yyyy-mm-dd (xx) | xxxxxxxxxxxx/ yyyy-mm-dd (xx) |
| xxxxxx | yyyy-mm-dd (xx) | xxxxxxxxxxxx/ yyyy-mm-dd (xx) |
| xxxxxx | yyyy-mm-dd (xx) | xxxxxxxxxxxx/ yyyy-mm-dd (xx) |
| Source: \\xx\xxx\xxx\xxx\xxx\xxxx\xx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | |

Programming Note: Sort by Treatment, Subject ID.

Listing 16.2.8.1 Hematology

Treatment: GLS-1200, Placebo

| Subject ID | Visit | Date/Time<br>(Study Day) | Lab Test | Result | Reference Range |
|---|---|---|---|---|---|
| xxxxxx | Day 0 | yyyy-mm-dd hh:mm (xx) | xxxxxxxxx | xx.x L, CS | xxxx - xxxx |
| | | | xxxxxxxxx | xx.x | xxxx - xxxx |
| | | | xxxxxxxxx | xx.x | xxxx - xxxx |
| | | | xxxxxxxxx | xx.x | xxxx - xxxx |
| | | | xxxxxxxxx | xx.x H, NCS | xxxx - xxxx |
| | | | xxxxxxxxx | xx.x | xxxx - xxxx |
| | | | xxxxxxxxx | xx.x | XXXX - XXXX |
| | | | XXXXXXXXX | XX.X | xxxx - xxxx |
| | Visit 4 | yyyy-mm-dd hh:mm (xx) | XXXXXXXXX | XX.X | XXXX - XXXX |
| | | | xxxxxxxxx | XX.X | xxxx - xxxx |

L=Low, H=High, (N)CS=(Not) Clinically Significant

date time

Programming Note: Repeat for Listing 16.2.8.2 Chemistry

Listing 16.2.8.3 Vital Signs

Treatment: GLS-1200, Placebo

| Subject ID Visit | Date/Time<br>(Study Day) | Diastolic Blood<br>Pressure<br>(mmHg) | Systolic Blood<br>Pressure<br>(mmHg) | Heart Rate<br>(beats/min) | Temperature<br>(C) | Height<br>(cm) | Weight<br>(kg) |
|---|---|---|---|---|---|---|---|
| xxxxxx Day 0<br>Week 2<br>Week 4<br>Week 6 | yyyy-mm-dd hh:mm (xx)<br>yyyy-mm-dd hh:mm (xx)<br>yyyy-mm-dd hh:mm (xx)<br>yyyy-mm-dd hh:mm (xx) | xx.x<br>xx.x<br>xx.x<br>xx.x | xx.x<br>xx.x<br>xx.x<br>xx.x | xx.x<br>xx.x<br>xx.x<br>xx.x | XX.X<br>XX.X<br>XX.X<br>XX.X | xx.x | xx.x |

date time

Protocol: T2R-002

#### Listing 16.2.8.4 12-Lead Electrocardiogram


Treatment: GLS-1200, Placebo

| Subject ID | Visit | ECG Date/Time<br>(Study Day) | Parameter | Result | Overall Interpretation | Abnormal Findings |
|---|---|---|---|---|---|---|
| XXXXXX | Day 0 | yyyy-mm-dd hh:mm (xx) | xxxxxxxxxxx | xx.x | Normal/Abnormal NCS/Abnormal CS | xxxxxxxxxxxxxxx |
| | | | XXXXXXXXXXX | XX.X | | |
| | | | XXXXXXXXXXX | XX.X | | |
| | | | XXXXXXXXXXX | xx.x | | |
| | | | XXXXXXXXXXX | XX.X | | |
| | | | XXXXXXXXXXX | xx.x | | |
| | | | XXXXXXXXXXX | xx.x | | |
| | | | XXXXXXXXXXX | xx.x | | |
| | Week 4 | yyyy-mm-dd hh:mm (xx) | xxxxxxxxxxx | xx.x | Normal/Abnormal NCS/Abnormal CS | xxxxxxxxxxxxxx |
| | | | xxxxxxxxxx | xx.x | | |
| | | | XXXXXXXXXXX | XX.X | | |
| | | | XXXXXXXXXXX | XX.X | | |
| | | | XXXXXXXXXXX | XX.X | | |
| | | | XXXXXXXXXXX | xx.x | | |
| | | | XXXXXXXXXXX | xx.x | | |
| | | | XXXXXXXXXXX | xx.x | | |

N(CS)=(Not) Clinically Significant

date

time

Listing 16.2.8.5 Physical Examination

Treatment: GLS-1200, Placebo

| Subject ID | Visit | Date | Exam | Clinically Significant Findings |
|---|---|---|---|---|
| | | (Study Day) | Performed | |
| xxxxxx | Day 0 | yyyy-mm-dd (xx) | Yes/No | Yes/No |
| | Week 2 | yyyy-mm-dd (xx) | Yes/No | Yes/No |
| | Week 4 | yyyy-mm-dd (xx) | Yes/No | Yes/No |
| | Week 6 | yyyy-mm-dd (xx) | Yes/No | Yes/No |
| xxxxxx | Day 0 | yyyy-mm-dd (xx) | Yes/No | Yes/No |
| | Week 2 | yyyy-mm-dd (xx) | Yes/No | Yes/No |
| | Week 4 | yyyy-mm-dd (xx) | Yes/No | Yes/No |
| | Week 6 | yyyy-mm-dd (xx) | Yes/No | Yes/No |

date

time

Listing 16.2.8.6 Pregnancy Test

Treatment: GLS-1200, Placebo

| Subject ID | Visit | Date<br>(Study Day) | Test Performed | Result |
|---|---|---|---|---|
| | | (Study Day) | | |
| xxxxxx | Day 0 | yyyy-mm-dd (xx) | Yes/No | Negative/Positive |
| | Week 2 | yyyy-mm-dd (xx) | Yes/No | Negative/Positive |
| | Week 4 | yyyy-mm-dd (xx) | Yes/No | Negative/Positive |
| xxxxxx | Day 0 | yyyy-mm-dd (xx) | Yes/No | Negative/Positive |
| | Week 2 | yyyy-mm-dd (xx) | Yes/No | Negative/Positive |
| | Week 4 | yyyy-mm-dd (xx) | Yes/No | Negative/Positive |

date time

## **DocuSign**

#### **Certificate Of Completion**

Envelope Id: 067D38AAE50F442C8CF9E1EEE7672DB4

Subject: Please DocuSign: GeneOne\_T2R-002\_SAP\_v2.0\_21JAN2022\_final.docx

Source Envelope:

Document Pages: 69 Certificate Pages: 5

AutoNav: Enabled

**Envelopeld Stamping: Disabled** 

Time Zone: (UTC-05:00) Eastern Time (US & Canada)

Status: Completed

Envelope Originator: Ahmed Tariq 5826 Fayetville Rd

Suite 202

Durham, NC 27713

ahmed.tariq@catalystcr.com IP Address: 67.86.44.161

#### **Record Tracking**

Status: Original

1/21/2022 2:43:50 PM

Holder: Ahmed Tariq

Signatures: 3

Initials: 0

ahmed.tariq@catalystcr.com

## Timestamp

Location: DocuSign

Sent: 1/21/2022 2:47:14 PM Viewed: 1/21/2022 2:47:50 PM Signed: 1/21/2022 2:48:43 PM

Sent: 1/21/2022 3:33:52 PM

Viewed: 1/21/2022 3:47:44 PM

Signed: 1/21/2022 3:48:48 PM

#### Signer Events

Ahmed Tariq

ahmed.tariq@catalystcr.com

Catalyst Clinical Research - Part 11

Security Level: Email, Account Authentication

(Required)

Ahmed Tarig

Signature ID:

Signature

8A9AFFC7-511B-4804-9134-C7E9728C3D84

Signature Adoption: Pre-selected Style

Using IP Address: 67.86.44.161

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

#### **Electronic Record and Signature Disclosure:**

Not Offered via DocuSign

Joel Maslow jmaslow@genels.us

Security Level: Email, Account Authentication

(Required)

DocuSigned by:

Joel Maslow

Signer Name: Joel Maslow Signing Reason: I approve this document Signing Time: 21-Jan-2022 | 12:48:44 PM PST -04EA2860227C41CB95FDE4D9283AF2C9

Signature Adoption: Pre-selected Style

Signature ID:

04EA2860-227C-41CB-95FD-E4D9283AF2C9

Using IP Address: 71.25.109.173

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

#### **Electronic Record and Signature Disclosure:**

Accepted: 1/21/2022 3:47:44 PM

ID: fb122045-6f6b-4297-9385-b5fe167eca46

| Signer Events | Signature | Timestamp |
|---|---|---|
| Susan E. Spruill | | Sent: 1/21/2022 2:47:15 PM |
| sspruill@appstatsconsulting.com | Susan E. Spruill | Viewed: 1/21/2022 5:06:49 PM |
| Security Level: Email, Account Authentication (Required) | | Signed: 1/21/2022 5:07:56 PM |
| | Signature Adoption: Pre-selected Style | |
| | Signature ID: | |
| | 6B44CB45-B795-4FD5-B700-ED25E98AB084 | |
| | Using IP Address: 99.197.222.18 | |
| | With Signing Authentication via DocuSign password | 1 |
| | With Signing Reasons (on each tab): | |
| | I approve this document | |

# Electronic Record and Signature Disclosure: Accepted: 1/21/2022 5:06:49 PM ID: d33f3acd-59af-4d13-a931-eeea026d5ce7

| <b>Electronic Record and Signature Discl</b> | osure | |
|---|---|---|
| Payment Events | Status | Timestamps |
| Envelope Sent Certified Delivered Signing Complete Completed | Hashed/Encrypted Security Checked Security Checked Security Checked | 1/21/2022 2:47:15 PM<br>1/21/2022 5:06:49 PM<br>1/21/2022 5:07:56 PM<br>1/21/2022 5:07:56 PM |
| Envelope Summary Events | Status | Timestamps |
| Notary Events | Signature | Timestamp |
| Witness Events | Signature | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Editor Delivery Events | Status | Timestamp |
| In Person Signer Events | Signature | Timestamp |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Catalyst Clinical Research - Part 11 (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

#### Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

#### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

#### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us

#### All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

#### **How to contact Catalyst Clinical Research - Part 11:**

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: shawnegerton@catalystcr.com

#### To advise Catalyst Clinical Research - Part 11 of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at shawnegerton@catalystcr.com and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

#### To request paper copies from Catalyst Clinical Research - Part 11

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to shawnegerton@catalystcr.com and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

#### To withdraw your consent with Catalyst Clinical Research - Part 11

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to shawnegerton@catalystcr.com and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

#### Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

#### Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify Catalyst Clinical Research Part 11 as described above, you consent to receive exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you by Catalyst Clinical Research Part 11 during the course of your relationship with Catalyst Clinical Research Part 11.